CLINICAL TRIAL: NCT01886729
Title: Effect of Time Shift of Transcranial Direct Current Stimulation (tDCS) for Treatment of Acute Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Sarah Rabau, University Hospital, Antwerp
Allocation: Randomized | Masking: None
Other Study IDs: EC 11/18/146
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Tinnitus
Keywords: transcranial direct current stimulation; time shift
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

ARMS (2):
- tDCS simultaneously with hyperbaric oxygen therapy (Active Comparator)
  Interventions: Other: transcranial direct current stimulation (tDCS)
- tDCS 3 weeks after start tinnitus (Active Comparator)
  Interventions: Other: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Other: transcranial direct current stimulation (tDCS)

SUMMARY:
The treatment for patients with acute tinnitus consists of Methylprednisolone and hyperbaric oxygen therapy. For this study transcranial direct current stimulation (tDCS) was added to the protocol. The purpose is to determine the effect of the time shift of tDCS. Two conditions will be compared: tDCS simultaneously with the hyperbaric oxygen therapy or tDCS 3 weeks after the start of the tinnitus.

An audiological testing will be performed at the day of admission, after 3 weeks, 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years
* presence of acute tinnitus or worsening of tinnitus caused by otogenic disease
* registration in UZA within 48 hours after start tinnitus
* VAS-score ≥ 4
* ability to understand and sign informed consent

Exclusion Criteria:

* history of epileptic seizures
* severe organic comorbidity
* psychiatric disorders or a history of psychiatric disorders with psychotic symptoms
* Pace maker
* pregnancy

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Dates: Start 2012-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of tinnitus | 12 weeks
  Tinnitus Questionnaire, Visual Analog Scale, Beck Depression Index, Hyperacusis questionnaire

SECONDARY OUTCOMES:
Hearing | 12 weeks
  Audiometry, Otoacoustic emissions, Tympanometry, Speech in noise

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Antwerp, Edegem, Antwerp, Belgium